CLINICAL TRIAL: NCT03496623
Title: A Phase 3, Randomized, Placebo-controlled, Double-blind, Adaptive Study to Evaluate the Safety and Efficacy of Inhaled Treprostinil in Patients With Pulmonary Hypertension Due to Chronic Obstructive Pulmonary Disease (PH-COPD)
Brief Title: A Phase 3 Adaptive Study to Evaluate the Safety and Efficacy of Inhaled Treprostinil in Participants With Pulmonary Hypertension (PH) Due to Chronic Obstructive Pulmonary Disease (COPD)
Acronym: PERFECT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIN-PH-304
Record Dates: First submitted 2018-03-29; First posted 2018-04-12 (Actual); Results first posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Hypertension; Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary Hypertension; COPD; Inhaled Treprostinil; 6-Minute Walk Test; Tyvaso
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inhaled Treprostinil (Experimental): Inhaled treprostinil delivered via an ultrasonic nebulizer with a target dosing regimen of 12 breaths (72 micrograms [mcg]) 4 times daily (QID)
  Interventions: Drug: Inhaled treprostinil solution
- Placebo (Placebo Comparator): Placebo delivered via an ultrasonic nebulizer for QID administration
  Interventions: Drug: Placebo solution

INTERVENTIONS:
Drug: Inhaled treprostinil solution — Treprostinil inhalation solution
  Arms: Inhaled Treprostinil
Drug: Placebo solution — Placebo solution
  Arms: Placebo

SUMMARY:
The primary objective of this study is to demonstrate the efficacy of inhaled treprostinil compared to placebo in improving exercise ability as measured by change from baseline in 6-Minute Walk Distance (6MWD) following 12 weeks of active treatment in participants with PH-COPD.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, 34-week, cross-over study, with a Treatment Period of approximately 26 weeks under the Original Crossover Design or, if applicable, a 21-week parallel study, with a Treatment Period of approximately 14 weeks under the Contingent Parallel Design.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet the following criteria may be included in the study:

1. Participant voluntarily gives informed consent to participate in the study.
2. Males and females 18 years of age and above at the time of informed consent.

   1. Women of childbearing potential (defined as less than 1 year post-menopausal and not surgically sterile) must agree to practice abstinence or use 2 highly effective methods of contraception (defined as a method of birth control that results in a low failure rate, [<1% per year], such as approved hormonal contraceptives, barrier methods [such as condom or diaphragm] used with a spermicide, or an intrauterine device) for the duration of study treatment and for 48 hours after discontinuing study drug. Participants must have a negative pregnancy test at the Screening Visit 1 (urine [prior to the first dose of study medication] and serum) and Baseline Visit (Study Week 1) (urine).
   2. Males with a partner of childbearing potential must agree to use a barrier method (condom) with a spermicide for the duration of treatment and for at least 48 hours after discontinuing study drug.
3. Diagnosis of PH-COPD (World Heath Organization [WHO] Group 3).
4. Clinical diagnosis of COPD will be made using the Global Initiative for Chronic

   Obstructive Lung Disease (GOLD) diagnostic criteria (GOLD Criteria 2020) and spirometry with the following documented parameters measured during Screening Visit 1 (prior to start of low-dose inhaled treprostinil):
   1. Forced expiratory volume in 1 second (FEV1) <80% predicted
   2. FEV1/Forced vital capacity (FVC) <70
5. The participant has a resting saturation peripheral capillary oxygenation (SpO2) greater than or equal to 90%, with or without supplemental oxygen, but not to exceed 10 liters (L)/min oxygen supplementation by any mode of delivery during Screening Visit 1.
6. During Screening Visit 1 prior to start of low-dose inhaled treprostinil, a 6MWD greater than or equal to 100 meters.
7. Have a right heart catheterization (RHC) performed during Screening Visit 1. (A previous RHC obtained within 12 months prior to the start of Screening Visit 1 is acceptable for determining eligibility, even if done without oxygen or vasodilator challenge, and a repeat RHC is not required.) The following parameters must be documented for eligibility:

   1. Pulmonary vascular resistance (PVR) greater than or equal to 4 Wood units
   2. A pulmonary artery wedge pressure (PAWP) or left ventricular end-diastolic pressure (LVEDP) of less than or equal to 15 millimeters of mercury (mmHg)
   3. A Pulmonary artery pressure mean (PAPm) of greater than or equal to 30 mmHg
8. Participants must be on a stable and optimized dose of chronic COPD medications for greater than or equal to 30 days prior to start of Screening Visit 1 and remain on the same dose throughout the Screening Period.
9. In the opinion of the Investigator, the participant can communicate effectively with study personnel and is considered reliable, willing, and likely to be cooperative with protocol requirements, including attending all study visits.

Exclusion Criteria:

The following will exclude participants from the study:

1. The participant has a diagnosis of either pulmonary arterial hypertension (PAH) or pulmonary hypertension (PH) due to reasons other than COPD. This would include, but is not limited to, chronic thromboembolic PH or acute/recent deep vein thrombosis or pulmonary embolism, untreated or inadequately treated obstructive sleep apnea, connective tissue disease (including but not limited to systemic sclerosis/scleroderma or systemic lupus erythematosus), sarcoidosis, human immunodeficiency virus-1 infection, and other conditions under WHO Group 1, 2, 4, and 5 classifications.
2. Based on chest computed tomography (CT) imaging during Screening Visit 1, the participant has a confirmed diagnosis of WHO Group 3 PH, other than COPD, such as idiopathic pulmonary fibrosis, combined pulmonary fibrosis and emphysema, diffuse parenchymal lung disease or interstitial lung disease. A previous chest CT scan performed within the 6 months prior to the start of Screening Visit 1 is also acceptable, and a repeat assessment is not required.

   A redacted CT scan report (from Screening Visit 1 or dated within prior 6 months) should be provided to the Medical Monitor with the Pre-Baseline Review Form to confirm eligibility.
3. The participant has received any Food and Drug Administration (FDA)-approved medication for the treatment of PAH (that is, prostacyclin, prostacyclin receptor agonist, endothelin receptor antagonist [ERA], phosphodiesterase type 5 inhibitor [PDE5-I], or soluble guanylate cyclase [sGC] stimulator) at Screening Visit 1 and thereafter, except if received for acute vasoreactivity testing.
4. The participant has a previous diagnosis of homozygous alpha-1 antitrypsin deficiency.
5. The participant has any prior intolerance to inhaled prostanoid therapy.
6. Inability to tolerate low-dose (3 breaths, 18 mcg) study drug and/or inability to follow dosing regimen during the Screening Period (pre-randomization).
7. Unwilling or unable to use Sponsor-provided devices (actigraph, spirometer, or smart device).
8. The participant has evidence of clinically significant left-sided heart disease (including but not limited to left ventricular ejection fraction <40%, left ventricular hypertrophy,) or clinically significant cardiologic conditions, such as congestive heart failure, coronary artery disease, or valvular heart disease. Note: Participants with abnormal left ventricular function attributable to the effects of right ventricular overload will not be excluded, but a discussion with and approval by the Sponsor Medical Monitor is needed.
9. Any exacerbation of COPD (including hospitalization or outpatient therapy) or active pulmonary or upper respiratory infection 60 days prior to start of Screening Visit 1 through the Baseline Visit. This is defined as worsening of respiratory symptoms that required treatment with corticosteroids and/or antibiotics.
10. Initiation of pulmonary rehabilitation within 12 weeks prior to start of Screening Visit 1 or, in the opinion of the Investigator, pulmonary rehabilitation is likely to be needed during the study Treatment Period.
11. The participant has any form of congenital heart disease (repaired or unrepaired; other than a patent foramen ovale).
12. The participant has any musculoskeletal disorder (severe arthritis of the lower limbs which limits ambulation, recent hip or knee joint replacement, artificial leg) or any other condition that would likely be the primary limitation to ambulation.
13. Use of any other investigational drug or device within 30 days prior to the start of Screening Visit 1.
14. Any other clinically significant illness or abnormal laboratory value(s) measured during the Screening Period that, in the opinion of the Investigator, might adversely affect the interpretation of the study data or safety of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — United Therapeutics
Locations (76):
- United States (65):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University Medical Center, Phoenix, Arizona
  - University of Arizona Clinical and Translational Science (CATS) Research Center, Tucson, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - Santa Barbara Pulmonary Associates, Santa Barbara, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - South Denver Cardiology, Littleton, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - St. Francis Medical Institute, Clearwater, Florida
  - University of Florida Clinical Research Center, Gainesville, Florida
  - St. Vincent's Lung, Sleep, and Critical Care Specialists, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Pulmonary Disease Specialists, Kissimmee, Florida
  - University of Miami Hospital, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Pulmonary & Critical Care of Atlanta, Atlanta, Georgia
  - Georgia Clinical Research, Austell, Georgia
  - University of Illinois Medical Center, Chicago, Illinois
  - Advocate Aurora Health Care, Elmhurst, Illinois
  - Advocate Condell Medical Center, Libertyville, Illinois
  - Advocate Heart Institute & Pulmonology, Normal, Illinois
  - Edward Heart Hospital, Oakbrook Terrace, Illinois
  - Indiana University Healh North Hospital, Indianapolis, Indiana
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Louisville Research Foundation, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Detroit Medical Center Lung Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Beaumont Health, Troy, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - The University of New Mexico, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - The Mount Sinai Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Carl and Edyth Lindner Research Center at the Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Clinical Research Associates of Central PA, LLC, DuBois, Pennsylvania
  - Temple Lung Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center - Montefiore, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Statcare Pulmonary Consultants, Knoxville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Tech, El Paso, Texas
  - Clear Lake Specialties/Tranquility Research, Webster, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (6):
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - El Cruce Hospital, Buenos Aires
  - Fundacion Favaloro, Ciudad Autonoma Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Hospital Italiano de Cordoba, Córdoba
  - Centro Medico 21 de Diciembre, Santa Fe
- Israel (4):
  - Lady Davis Carmel Medical Centre, Haifa
  - Hadassah-Hebrew University Hospital, Jerusalem
  - Rabin Medical Center, Petah Tiva
  - The Chaim Sheba Medical Center, Tel Litwinsky
- CardioPulmonary Research Center, Guaynabo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nathan SD, Argula R, Trivieri MG, Aziz S, Gay E, Medarov B, Parambil J, Raina A, Risbano MG, Thenappan T, Soto JS, Bell H, Lacasse V, Sista P, Di Marino M, Smart A, Hawkes B, Nelson E, Bull T, Tapson V, Waxman A. Inhaled treprostinil in pulmonary hypertension associated with COPD: PERFECT study results. Eur Respir J. 2024 Jun 6;63(6):2400172. doi: 10.1183/13993003.00172-2024. Print 2024 Jun. PMID 38811045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 188 participants were enrolled; 80 of the 188 enrolled participants were screen failures prior to the Run-In Period. Per prespecified analysis, data were not collected for the participants who were screen failures.
Pre-assignment Details: In the Original Crossover Design, a total of 64 participants were randomized to 1 of 2 treatment sequences (treprostinil-placebo) or (placebo-treprostinil) in a crossover study design for 12 weeks during 2 dosing periods. There was a washout of at least 7 days between the dosing periods. 12 participants were randomized to receive either treprostinil or placebo during the single treatment period in Contingent Parallel Design.
Groups:
- Run-In: Participants received low dose treprostinil for inhalation for up to 2 weeks before randomization
- Original Crossover Design - Treprostinil, Then Placebo: Participants received either treprostinil or placebo in the following order:
  Period 1: Up to 72 micrograms (μg) of treprostinil for inhalation four times daily (QID), for up to 12 weeks Period 2: Placebo QID for up to 12 weeks
- Original Crossover Design - Placebo, Then Treprostinil: Participants received either treprostinil or placebo in the following order:
  Period 1: Placebo QID for up to 12 weeks Period 2: Up to 72 μg of treprostinil for inhalation QID, for up to 12 weeks
- Contingent Parallel Design - Treprostinil: Participants received up to 72 μg of treprostinil for inhalation QID, for up to 12 weeks
- Contingent Parallel Design - Placebo: Participants received placebo to match treprostinil QID, for up to 12 weeks
Period: Run-In Period (2 Weeks)
Arm/Group | Run-In | Original Crossover Design - Treprostinil, Then Placebo | Original Crossover Design - Placebo, Then Treprostinil | Contingent Parallel Design - Treprostinil | Contingent Parallel Design - Placebo
Started | 108 | 0 | 0 | 0 | 0
Received At Least 1 Dose of Study Drug | 108 | 0 | 0 | 0 | 0
Completed | 76 | 0 | 0 | 0 | 0
Not Completed | 32 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Discontinued Prior to Randomization | 31 | 0 | 0 | 0 | 0
Period: Period 1 (12 Weeks)
Arm/Group | Run-In | Original Crossover Design - Treprostinil, Then Placebo | Original Crossover Design - Placebo, Then Treprostinil | Contingent Parallel Design - Treprostinil | Contingent Parallel Design - Placebo
Started | 0 (108 participants enrolled to receive a low dose of treprostinil for 2 weeks during safety Run-In (before randomization) as part of screening. Data for this cohort are only included in Mortality and Adverse Events.) | 32 | 32 | 6 | 6
Received At Least 1 Dose of Study Drug | 0 | 32 | 32 | 6 | 6
Completed | 0 | 26 | 29 | 5 | 4
Not Completed | 0 | 6 | 3 | 1 | 2
Not completed — Death | 0 | 3 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 3 | 0 | 0
Period: Period 2 (12 Weeks)
Arm/Group | Run-In | Original Crossover Design - Treprostinil, Then Placebo | Original Crossover Design - Placebo, Then Treprostinil | Contingent Parallel Design - Treprostinil | Contingent Parallel Design - Placebo
Started | 0 (108 participants enrolled to receive a low dose of treprostinil for 2 weeks during the safety Run-In (before randomization) as part of screening. Data for this cohort are only included in Mortality and Adverse Events.) | 26 | 29 | 0 (No participants were planned for Period 2 in this cohort) | 0 (No participants were planned for Period 2 in this cohort)
Received At Least 1 Dose of Study Drug | 0 | 20 | 28 | 0 | 0
Completed | 0 | 19 | 21 | 0 | 0
Not Completed | 0 | 7 | 8 | 0 | 0
Not completed — COVID-19 Pandemic Impact | 0 | 4 | 5 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all participants who were randomized and received at least one dose of study drug.
Groups:
- Original Crossover Design: Participants were randomized to one of two treatment sequences: treprostinil-placebo, or placebo-treprostinil during two dosing periods, each up to 12 weeks
- Total: Total of all reporting groups
Arm/Group | Original Crossover Design | Contingent Parallel Design - Treprostinil | Contingent Parallel Design - Placebo | Total
Number analyzed (Participants) | 64 | 6 | 6 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (7.83) | 70.3 (6.71) | 73.3 (2.16) | 69.7 (8.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 0 | 2 | 33
  Male | 33 | 6 | 4 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 4
  Not Hispanic or Latino | 62 | 6 | 4 | 72
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 1 | 2 | 18
  White | 47 | 5 | 4 | 56
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in 6-Minute Walk Distance (6MWD)
Description: 6 MWD was calculated at peak exposure (10 to 60 minutes after dosing). 6MWT was performed by standardized procedures for all participants. Participants were asked to walk a set course for 6 minutes (timed) and the distance walked (in meters) was recorded. Statistical analyses were not performed due to lack of appropriate sample size.
Time Frame: Baseline, Week 12
Population: Full Analysis Set included all participants who were randomized and received at least one dose of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure and 'Number analyzed' = participants evaluable at the specified timeframe.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Original Crossover Design - Treprostinil; Contingent Parallel Design - Treprostinil: Participants received up to 72 μg of treprostinil for inhalation QID, for up to 12 weeks
- Original Crossover Design - Placebo: Participants received placebo to match treprostinil for inhalation QID, for up to 12 weeks
Arm/Group | Original Crossover Design - Treprostinil | Original Crossover Design - Placebo | Contingent Parallel Design - Treprostinil | Contingent Parallel Design - Placebo
Number analyzed (Participants) | 46 | 47 | 6 | 5
meters
  Baseline | 225.07 (77.41) | 220.47 (77.64) | 231.50 (60.77) | 283.00 (67.78)
  Change at Week 12: number analyzed (Participants) | 38 | 42 | 3 | 4
  Change at Week 12 | -4.47 (39.01) | -5.14 (50.71) | 20.33 (116.99) | 18.5 (42.49)

2. Secondary Outcome: Change From Baseline to Week 12 in Moderate to Vigorous Physical Activity (MVPA)
Description: MVPA was defined as the number of minutes spent in moderate to vigorous physical activity as measured via a wrist-worn medical grade physical activity monitor. The screening data were used to establish a baseline level of physical activity.
Time Frame: Baseline, Week 12
Population: Full Analysis Set included all participants who were randomized and received at least one dose of study drug. Data were not collected for this outcome measure due to study termination and lack of appropriate sample size.
Groups:
- Original Crossover Design - Treprostinil; Contingent Parallel Design - Treprostinil: Participants received up to 72 μg of treprostinil for inhalation four times daily, for up to 12 weeks
- Original Crossover Design - Placebo: Participants received placebo to match treprostinil for inhalation four times daily, for up to 12 weeks
- Contingent Parallel Design - Placebo: Participants received placebo to match treprostinil four times daily, for up to 12 weeks
Arm/Group | Original Crossover Design - Treprostinil | Original Crossover Design - Placebo | Contingent Parallel Design - Treprostinil | Contingent Parallel Design - Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline to Week 12 in Overall Activity
Description: Overall activity was defined as the number of minutes spent in overall activity (non-sedentary activity) as measured via a wrist-worn medical grade physical activity monitor. The screening data will be used to establish a baseline level of physical activity.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Arm/Group | Original Crossover Design - Treprostinil | Original Crossover Design - Placebo | Contingent Parallel Design - Treprostinil | Contingent Parallel Design - Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline to Week 12 in Borg Dyspnea Score
Description: The Borg Dyspnea Score was a 11-point scale rating the maximum level of dyspnea experienced during the 6-minute walking test (6MWT). Scores range from 0 (no dyspnea at all) to 10 (very, very severe dyspnea), with lower scores indicating a less exertion (a better outcome). The Borg Dyspnea Score was to be evaluated immediately after the 6MWT.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Arm/Group | Original Crossover Design - Treprostinil | Original Crossover Design - Placebo | Contingent Parallel Design - Treprostinil | Contingent Parallel Design - Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline to Week 12 in 6MWD/Borg Dyspnea Composite Score
Description: 6MWD was calculated at peak exposure (10 to 60 minutes after dosing). 6MWT was performed by standardized procedures for all participants. Participants were asked to walk a set course for 6 minutes (timed) and the distance walked (in meters) was recorded. The Borg Dyspnea Score was an 11-point scale rating the maximum level of dyspnea experienced during the 6MWT. Scores range from 0 (no dyspnea at all) to 10 (very, very severe dyspnea), with lower scores indicating less exertion (a better outcome). The Borg Dyspnea Score was to be evaluated immediately after the 6MWT. The average 6WMWD data and the average Borg Dyspnea Composite Score data were summed and reported as the composite score.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Arm/Group | Original Crossover Design - Treprostinil | Original Crossover Design - Placebo | Contingent Parallel Design - Treprostinil | Contingent Parallel Design - Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline to Week 12 in Quality of Life (QOL) Measured by St. George's Respiratory Questionnaire (SGRQ)
Description: The SGRQ is a designed to measure how breathing impacts overall health, daily life, and perceived well-being in participants with obstructive airways disease. Scores range from 0 to 100, with lower scores indicating a better QoL.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Arm/Group | Original Crossover Design - Treprostinil | Original Crossover Design - Placebo | Contingent Parallel Design - Treprostinil | Contingent Parallel Design - Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline to Week 12 in QOL Measured by the University of California San Diego Shortness of Breath Questionnaire (UCSD SOBQ)
Description: The UCSD SOBQ is a self-administered rating of dyspnea associated with activities of daily living. The questionnaire uses a 6-point scale where 0 = "not at all" and 5 = "maximal or unable to do because of breathlessness". Lower scores indicate a better QoL.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Arm/Group | Original Crossover Design - Treprostinil | Original Crossover Design - Placebo | Contingent Parallel Design - Treprostinil | Contingent Parallel Design - Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline to Week 12 in Plasma Concentration of N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) Levels
Description: The NT-proBNP concentration is a biomarker associated with changes in right heart morphology and function. Improvement is defined as a decrease in the NT-proBNP plasma concentration.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Arm/Group | Original Crossover Design - Treprostinil | Original Crossover Design - Placebo | Contingent Parallel Design - Treprostinil | Contingent Parallel Design - Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline to Week 12 in Patient Global Assessment (PGA)
Description: The PGA is used to rate participant fatigue and shortness of breath. Participants will use the Sponsor-provided smart device for at-home capture of PGA data. The PGA used a 5-point response scale of: "never," "rarely," "sometimes," "often," or "always" with higher scores indicating a worse symptom rating.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Arm/Group | Original Crossover Design - Treprostinil | Original Crossover Design - Placebo | Contingent Parallel Design - Treprostinil | Contingent Parallel Design - Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Safety Analysis Set included all participants who received at least one dose of study drug. Data were prespecified to be collected by the treatment received for both treprostinil or placebo regardless of whether the treatment was received during the Original Crossover Design or the Contingent Parallel Design. Number of deaths that led to study discontinuation are reported in Participant Flow and number of deaths due to All-Cause Mortality are reported below.
Groups:
- Treprostinil: Participants who received up to 72 μg of treprostinil for inhalation QID, for up to 12 weeks during both the original cross-over design and the contingent parallel design combined
- Placebo: Participants who received placebo to match treprostinil QID, for up to 12 weeks during both the original cross-over design and the contingent parallel design combined
Arm/Group | Run-In | Treprostinil | Placebo
All-Cause Mortality (participants affected / at risk) | 1/108 | 5/66 | 0/58
Serious Adverse Events (participants affected / at risk) | 9/108 | 17/66 | 6/58
Other Adverse Events (participants affected / at risk) | 50/108 | 36/66 | 25/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In (N=108) | Treprostinil (N=66) | Placebo (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Brain injury (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In (N=108) | Treprostinil (N=66) | Placebo (N=58)
Fatigue (General disorders) | 2 | 7 | 2
Chest discomfort (General disorders) | 3 | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Headache (Nervous system disorders) | 9 | 7 | 4
Dizziness (Nervous system disorders) | 2 | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 19 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 11 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3

LIMITATIONS AND CAVEATS:
Per sponsor decision, the study was terminated early. Data were not collected for the secondary outcome measures due to study termination and lack of appropriate sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution clinical trial centers and PIs agreed not to publish or publicly present any results of clinical trial without prior written consent of sponsor, not to be withheld or delayed except as necessary to require removal of any sponsor confidential information (other than as necessary to fully disclose the trial design and results in accordance with applicable publication standards) or as necessary to provide reasonable time for sponsor to perfect any arising intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT03496623/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT03496623/SAP_001.pdf